CLINICAL TRIAL: NCT03014193
Title: Simplifying First Trimester Medical Abortion Follow-up
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 6009
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Medical Abortion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: Semiquantitative Multi-Level Pregnancy Test

SUMMARY:
This study evaluates the usability of the multilevel pregnancy test among women undergoing medical abortion.

ELIGIBILITY:
Inclusion Criteria:

* Have a first trimester pregnancy with a gestational age of ≤63 days;
* Desire medical abortion with mifepristone and misoprostol and be medically eligible for that treatment, according to clinic protocol;
* Be able to read and understand the local language or Russian;
* Have access to a telephone;
* Agree to follow all study procedures;
* Have no contraindication to participation in the study, in the judgment of the site investigator or designee.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women seeking medical abortion with pregnancies of 63 days or less.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Understanding of the instructions for the multilevel pregnancy test | 14 days
Ability to independently use the multilevel pregnancy tests | 14 days
Ability to interpret the results of the multilevel pregnancy test | 14 days

CONTACTS AND LOCATIONS:
Locations (5):
- Armenia (2):
  - Gyumri Maternity Hospital, Gyumri
  - Republican Institute of Reproductive Health, Perinatology, Obstetrics and Gynecology, Yerevan
- Georgia (2):
  - Batumi International Hospital, Batumi
  - David Gagua Clinic, Tbilisi
- City Policlinic #17, Almaty, Kazakhstan